CLINICAL TRIAL: NCT02763280
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Ginseng Extract on Improvement of Bone Metabolism in Menopausal Women
Brief Title: Efficacy and Safety of Ginseng Extract on Improvement of Bone Metabolism in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RDA-BM-GE
Record Dates: First submitted 2016-03-09; First posted 2016-05-05 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ginseng extract 1g (Experimental): Ginseng extract 1g
  Interventions: Dietary Supplement: Ginseng extract 1g
- Ginseng extract 3g (Experimental): Ginseng extract 3g
  Interventions: Dietary Supplement: Ginseng extract 3g
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginseng extract 1g — Ginseng extract 1g, parallel design
  Arms: Ginseng extract 1g
Dietary Supplement: Ginseng extract 3g — Ginseng extract 3g, parallel design
  Arms: Ginseng extract 3g
Dietary Supplement: Placebo — placebo, parallel design
  Arms: Placebo

SUMMARY:
Recently, osteoporosis has been recognized as a serious health problem in the elderly, it has also increased in young • middle-aged layer. Ginseng is history 2, 000 years Korean typical herbal medicine which is used as a medicinal is known the mystery of Elixir from a long time ago. A previous study was administered ginseng extract results in animal models induced osteoporosis, the bone-related biomarkers, including improved bone density and bone mass.

DETAILED DESCRIPTION:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of ginseng extract on improvement of Bone metabolism in menopausal women. The investigators measured Serum Osteocalcin, Urinary Deoxypyridinoline, DPD/OC ratio, Serum CTX, NTX, Ca, Phosphorus, BSALP(vone specific-alkaline phosphatase), P1NP(Procollagen type 1 N-terminal propeptide), WOMAC index(Western Ontario and McMaster Universities Arthritis).

ELIGIBILITY:
Inclusion Criteria:

* age older than 40 years, after a amenorrhea 6 months in women
* T-score less than -1.0,
* osteocalcin 8(ng/mL) or more and DPD 5.2(nMDPD/mMcreatinine) or more,
* subjects giving written informed consent

Exclusion Criteria:

* Diagnosed osteoporosis
* BMI ≤ 18.5kg/m2 or BMI ≥ 30 kg/m2
* Cardiovascular disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnancy or breast feeding etc,.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in Serum Osteocalcin | Baseline and 12 week
  Serum Osteocalcin was measured in study baseline and visit 3(12 week).
Changes in Urinary Deoxypyridinoline | Baseline and 12 week
  Urinary Deoxypyridinoline was measured in study baseline and visit 3(12 week).
Changes in DPD/OC ratio | Baseline and 12 week
  DPD/OC ratio was measured in study baseline and visit 3(12 week)

SECONDARY OUTCOMES:
Changes in Serum CTX(Cross-linked C-telopeptide of type-1 collagen) | Baseline and 12 week
  Serum CTX was measured in study baseline and visit 3(12 week)
Changes in Serum NTX(Cross-linked N-telopeptide of type-1 collagen) | Baseline and 12 week
  Serum NTX was measured in study baseline and visit 3(12 week)
Changes in Serum Ca, Phosphorus | Baseline and 12 week
  Serum Ca, Phosphorus was measured in study baseline and visit 3(12 week)
Changes in Serum BSALP(bone specific-alkaline phosphatase) | Baseline and 12 week
  Serum BSALP was measured in study baseline and visit 3(12 week)
Changes in Serum P1NP(procollagen type 1 N-terminal propeptide) | Baseline and 12 week
  Serum P1NP was measured in study baseline and visit 3(12 week)
Changes in WOMAC index(Western ontario and mcmaster universities arthritis) | Baseline and 12 week
  WOMAC index was measured in study baseline and visit 3(12 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea